CLINICAL TRIAL: NCT02784184
Title: COPENHAGEN Minipuberty Study
Acronym: CPHMINIPUB
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anders Juul, Anders Juul, MD, PhD, DmSc, Rigshospitalet, Denmark
Other Study IDs: RH-H-15014876; RH-2015-210-04146 (Other: Danish Data Protection Agency)
Record Dates: First submitted 2016-05-17; First posted 2016-05-27 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Child Development; Disorders of Sex Development
Keywords: Hypothalamic-pituitary-gonadal axis
MeSH Terms: conditions — Disorders of Sex Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA EDTA-Blood Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 year follow-up group: 1 year follow-up group including 6 measurements
- 40 days diaper study subgroup: Subgroup of the "1 year follow-up group" including 15 girls undergoing daily measurement of urinary hormone excretion

SUMMARY:
Minipuberty is a term used to describe the transient activation of the pituitary-gonadal axis 2-3 months after birth in both boys and girls. It is, however, not known why infants reach adult levels of reproductive hormones in early life, nor is the exact timing of the peak known. Furthermore, what determines the timing of peaks and suppressions of reproductive hormones from infancy throughout childhood and into adolescence remains to be elucidated.

The study aims to described and evaluate dynamic changes in the hypothalamic-pituitary- gonadal axis in early postnatal life.

DETAILED DESCRIPTION:
Minipuberty is a term used to describe the transient activation of the pituitary-gonadal axis 2-3 months after birth in both boys and girls. It is, however, not known why infants reach adult levels of reproductive hormones in early life, nor is the exact timing of the peak known. Furthermore, what determines the timing of peaks and suppressions of reproductive hormones from infancy throughout childhood and into adolescence remains to be elucidated.

Few studies have investigated minipuberty and one, for example, found that it is affected in premature infants (before gestation week 37). However, no studies on normative data throughout minipuberty in infants exist.

Furthermore, using minipuberty as a window for diagnosis of endocrine disorders and future reproductive function has been suggested. Defining minipuberty, both in terms of circulating hormone levels and urinary metabolites, in healthy infants is therefore essential in order to utilize this window. Studies using patients with Disorders of Sex Development during minipuberty have been carried out, but they are hampered by small sample sizes and lack of control groups.

In addition, little is known about the genetic and epigenetic factors that drive the onset, progression and termination of minipuberty as well as the actual puberty, i.e. the factors responsible for the quiescence of the HPG axis during childhood and the dis-inhibition responsible for pubertal onset. Therefore, much attention was drawn on the study performing whole exome sequencing in patients and relatives with central precocious puberty (CPP). For the first time, MKRN3 was suggested as the primary factor responsible for HPG inhibition during mid-childhood. A number of studies support that MKRN3 mutations cause CPP, and genetic variation of MKRN3 affect pubertal timing in healthy girls. Our findings of declining serum levels of MKRN3 prior to pubertal onset in healthy girls support MKRN3 as a regulator of pubertal onset. The exact mechanism through which MRKN3 exceeds its effect remains to be elucidated; however, its zink-finger structure indicates regulation of superior cellular processes such as epigenetic regulation of DNA transcription.

Twin studies suggest that 60% of the inter-individual variation is caused by genetic factors. However, genome wide association (GWA) studies only explain a fraction of the variation in age at puberty. Recently, our research group has revealed the largest effect of a single SNP on age at pubertal onset in girls. The location of the SNPs in genes regulating FSH action emphasizes the need of a wide focus including downstream processes in the HPG axis when evaluating factors regulating puberty.

In general, the abovementioned studies have led to a spark in the interest in epigenetic studies, i.e. studies of genetic changes that are not caused by changes in the DNA sequences themselves, but rather regulatory mechanisms of DNA expression. Generally, this is thought to include DNA methylation, histone modifications and small RNAs. Epi-mutations (improper epigenetic regulation) possibly account for more of the variation in puberty than genetic factors. Previously, both gene-specific and genome-wide DNA methylation patterns have been studied. Genome-wide hypomethylation seen in peripheral leukocytes has been shown to be linked with an array of cancers, including colorectal cancers. As multiple histone modifications exist and analysis requires special sample treatment procedures, DNA methylation is the most appropriate epigenetic marker to analyze. A study of rats found that specific gene hypomethylation was accountable for lack of pubertal onset, but the link between epigenetics and mini- and pubertal timing and progression has, however, only scarcely been studied. Understanding this link would greatly add to our knowledge of reproductive function and normal sex development.

Disorders of Sex Development (DSD) is an umbrella term covering conditions with congenital disordered development of chromosomal, gonadal or anatomical sex. Genital abnormalities may include as many as up to 4-6 in 1000 births, although individual disorders are much rarer, e.g. 45,X/46,XY mosaicism is seen in about 1 in 15000 live births. Previously DSD diagnoses were labeled with different and often imprecise terms such as 'intersex', 'sex reversal' and 'hermaphroditism' etc. In 2006, DSD nomenclature was renamed and grouped according to genetic sex into sex chromosome DSD, 46,XY DSD and 46,XX DSD.

DSD patients are diagnosed at different periods in life depending on their diagnosis, phenotype and primary and secondary sexual development. Patients with sex chromosome DSD can be diagnosed at prenatal screenings, patients with affected external genitalia at birth, some during childhood due to growth abnormalities, some during adolescence due to abnormal pubertal progression and lastly, some in adulthood due to infertility.

Understanding normal sex development is therefore the key to identifying and optimizing diagnosis and treatment of patients with DSD. A project, as the present, that seeks to investigate normal minipuberty while comparing to minipuberty in patients with DSD is therefore of great importance. Furthermore, knowledge of the genetic and epigenetic control mechanisms of minipuberty will aid the understanding of reproductive physiology and in particular DSD pathology.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Maternal and paternal Caucasian origin
* Maternal pre-pregnancy BMI between 18 and 35 kg/m2
* No serious maternal illness, including no pre-existing maternal diabetes nor thyroid gland diseases
* Term pregnancy (week 37+0 to 41+7)
* No gestational diabetes
* No fetal malformations or chromosomal disorders
* Birth weight of child between 3rd and 97th percentile

Only healthy infants born at term will be included in the study which all prospective participants will be informed of.

Exclusion Criteria:

-

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pregnant women, meeting the inclusion criteria, and the fathers-to-be followed at the Department of Obstetrics, Rigshospitalet. Further, parents and infants with disordered sexual development (DSD). These patients will be recruited via The Department of Growth and Reproduction, Rigshospitalet. Parents whose fetuses have been diagnosed prenatally with any DSD diagnosis or during the first 6 months of life will be invited to participate.
  Three groups of participants in this study:
  1. A group of healthy infants
  2. All infant patients diagnosed with or under evaluation for DSD
  3. The parents of the healthy infants and DSD patients
  Number (approximately) of participants:
  1. 200 healthy infants (100 boys and 100 girls)
  2. unknown number of DSD infants that will be referred within a year to the Department of Growth and Reproduction; estimation: 15 DSD infants.
  3. 400 parents of healthy infants (200 fathers and 200 mothers) - unknown number of parents of DSD patients
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Serum and urinary metabolites of reproductive hormones (e.g. steroid hormone metabolites and gonadotropins) (newborn) | 3-7d, and 1,3,5,7,12m or 2,4,6,8,12m after birth plus 40 days daily measurement (urine, female 40 days diaper study subgroup)
  change/course serum and urinary metabolites
Urinary metabolites of endocrine disrupting chemicals (e.g. phthalates, phenols, perfluorinated compounds and parabens) (newborn) | 3-7d, & 1,3,5,7,12m or 2,4,6,8,12m after birth plus 40 days daily measurement (urine, female 40 days diaper study subgroup)
  change/course urinary metabolites
Basic clinical examination (newborn) (size and proportions) | 3-7d, and 1,3,5,7,12m or 2,4,6,8,12m after birth
  change/course: measurements of length, weight, skin folds and hip-waist ratio
Basic clinical examination (newborn) (pubertal staging) | 3-7d, and 1,3,5,7,12m or 2,4,6,8,12m after birth
  change/course: pubertal staging using Tanners classification (including testicular size in boys assessed by Prader's orchidometer and ultrasound
Basic clinical examination (newborn) (genitalia) | 3-7d, and 1,3,5,7,12m or 2,4,6,8,12m after birth
  change/course: classification of external genitalia (classification of genital tubercle, location of gonads, position of urethra, labia/scrotal fusion)
Basic clinical examination (newborn) (penile measurement) | 3-7d, and 1,3,5,7,12m or 2,4,6,8,12m after birth
  change/course: penile measurement with a ruler (in boys)
Basic clinical examination (newborn) (AGD) | 3-7d, and 1,3,5,7,12m or 2,4,6,8,12m after birth
  change/course: ano-genital distance (AGD) measured with a ruler
Genetic profiling | single determination or 3-7d, and 1,3,5,7,12m or 2,4,6,8,12m after birth
  Genotyping of different genetic loci (genetic variation of loci regulating hormone signalling, e.g. FSHB, etc.)
Epigenetic profiling | single determination or 3-7d, and 1,3,5,7,12m or 2,4,6,8,12m after birth
  change/course: epigenetic variation of loci regulating hormone signalling

SECONDARY OUTCOMES:
Basic clinical examination (parents) (height) | postpartal (within first 3 months)
  Height
Basic clinical examination (parents) (weight) | postpartal (within first 3 months)
  self-reported pre-pregnancy weight for the mother and postpartal weight of the father
Basic clinical examination (parents) | postpartal (within first 3 months)
  Skinfolds measured above the biceps, triceps, at the flank, and below the scapula
Pregnancy and perinatal outcome (newborn and mother) | before birth and perinatal phase
  Perinatal outcome including birth weight, -length, partus mode, adverse events/complications, pre- and perinatal drug intake, pregnancy outcomes including gestational age, pregnancy complications, IVF Treatment etc.
Medical history and exposure (parents) (basic) | postpartal (within first year)
  Basic medical history (parents) (questionaire / journal)
Medical history and exposure (parents) (obstetrical) | postpartal (within first year)
  Obstetrical history including outcomes of previous pregnancies and births (mother), smoking and drug intake during pregnancy (mother) (questionaire / journal)
Medical history and exposure (parents) (puberty) | postpartal (within first year)
  Pubertal history (parents) including age at menarche, pubertal timing with regard to peers, age at menopause of the mother of the parents etc. (questionaire)
Breastfeeding and food intake (newborn) | first year of life
  change/course: breastfeeding and food intake of the newborn during the course of the first year (questionaire)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Juul, Prof., Study Chair — Rigshospitalet, Denmark; Alexander S Busch, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Growth and Reproduction, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ljubicic ML, Busch AS, Upners EN, Fischer MB, Petersen JH, Raket LL, Frederiksen H, Johannsen TH, Juul A, Hagen CP. A Biphasic Pattern of Reproductive Hormones in Healthy Female Infants: The COPENHAGEN Minipuberty Study. J Clin Endocrinol Metab. 2022 Aug 18;107(9):2598-2605. doi: 10.1210/clinem/dgac363. PMID 35704034
- [Derived] Ljubicic ML, Busch AS, Upners EN, Fischer MB, Main KM, Andersson AM, Johannsen TH, Hagen CP, Juul A. Dynamic changes in LH/FSH ratios in infants with normal sex development. Eur J Endocrinol. 2022 Jun 1;187(1):135-142. doi: 10.1530/EJE-21-0999. PMID 35521767